CLINICAL TRIAL: NCT03501576
Title: Evaluation of Human Immune Responses Vaccination in Patients With Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andres Chang, Principal Investigator, Emory University
Other Study IDs: IRB00101067; NCI-2017-02313 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4236-17 (Other: Winship Cancer Institute)
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, T-Cell | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Inactivated Influenza Vaccine: Patients will be vaccinated with an FDA approved seasonal inactivated influenza vaccine
  Interventions: Biological: Inactivated Influenza Vaccine
- Qualifying subjects to receive a SARS-CoV2 vaccine.: Patients receive a SARS-CoV2 vaccine.
- Clinical Group Receiving SARS-CoV2 Booster Vaccines: Patients receive a SARS-CoV2 vaccine.

INTERVENTIONS:
Biological: Inactivated Influenza Vaccine — Given seasonal inactivated influenza vaccine IM
  Other Names: Fluzone Quadrivalent; Fluzone Quadrivalent Influenza Vaccine; Quadrivalent Influenza Vaccine; Quadrivalent Inactivated Influenza Vaccine; Flu Vaccine
  Groups: Inactivated Influenza Vaccine

SUMMARY:
This clinical trial evaluates the influenza virus vaccination in evaluating human immune response in patients with lymphoma. Evaluating immune response may increase the understanding of how the immune system changes when patients receive treatment for lymphomas by looking at the antibody levels and the level of the different cells that make up the immune system over time compared to those without lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the seroprotection and seroconversion rates after influenza or SARS-CoV2 vaccination in patients with lymphoma receiving active treatment or in follow up observation.

SECONDARY OBJECTIVES:

I. To characterize virus-specific plasmablasts and memory B cells after vaccination in patients with lymphoma receiving active treatment or in follow up observation.

II. To investigate the longevity of viral-specific humoral immunity to influenza virus in patients with lymphoma receiving active treatment or in follow up observation.

III. To assess the timing and strength of the peak immune response to vaccination.

IV. To assess the effect of different lymphomas and treatment modalities in the immune response to vaccination.

OUTLINE:

Patients receive seasonal inactivated influenza vaccine intramuscularly (IM) at day 0.

After completion of study treatment, patients are followed up at days 7, 28, 90, 180, and 365.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of lymphoma falling into the following categories:

  * B-NHL who have received 1 cycle of chemotherapy
  * B-NHL in complete remission and within 12 months after completion of chemotherapy
  * Chronic lymphocytic leukemia (CLL) or mantle cell lymphoma (MCL) receiving ibrutinib for at least 1 month
  * B-NHL in complete remission for over 12 months
  * Aggressive peripheral T-cell lymphoma (PTCL) who have received 1 cycle of chemotherapy
* Subject capable of providing written or electronic informed consent prior to initiation of any study procedures; subjects able to understand and comply with planned study procedures and be available for all study visits.

  * Screening labs must be within the following ranges or considered to be not clinically significant by the investigator:

Hematology:

* Hemoglobin: 7.0-16.1 gm/dL
* Platelet count: 10-600/µL
* Subjects who have not received the seasonal influenza vaccine in the current flu season and are not suspected to have had an influenza infection in the current flu season *- Platelet count: 10-600/uL

  * For cohort 1: Subjects who have not received the seasonal influenza vaccine in the current flu season and are not suspected to have had an influenza infection in the current flu season.
  * For cohort 3: Subjects must have previously received at least 1 dose of SARS-CoV2 vaccine. Patients who have not receive a prior SARS-CoV2 vaccine will be eligible to enroll in cohort.

Exclusion Criteria:

* Known infection with human immunodeficiency virus (HIV). This information will be obtained verbally from the patient
* Have any medical disease or condition that, in the opinion of the site principal investigator is a contraindication to study participation; this includes any chronic medical condition, defined as persisting 3 months (defined as 90 days) or longer, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject?s successful completion of this study
* Have an acute illness, as determined by the site principal investigator within 72 hours prior to study vaccination; an acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol and was not due to an influenza infection
* Subjects taking long-term systemic steroids defined as greater than 3 months in the past 12 months
* Have known hypersensitivity or allergy to eggs, egg or chicken protein, or other components of the study vaccine
* Have a history of Guillain-Barre syndrome (GBS)
* Subjects who had or are suspected to have had an influenza infection in the current influenza season
* Subjects who, at screening, have abnormal vital signs and/or physical exam, including a temperature ≥ 38.0 C, systolic blood pressure ≤ 90 or > 180 mmHg, pulse ≤ 60 or > 130 beats per minute, new rash, signs of infection
* Subjects who have already received the seasonal influenza vaccine in the current influenza vaccination season
* Subjects enrolled in hospice or whose life expectancy is less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients per observation group
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Percentage of subjects achieving seroprotection, defined as the percentage of subjects with a post-vaccination HI titer > 1:40 | Up to 180 days after immunization
  Rates of seroprotection will be calculated for each patient group, and 95% exact binomial confidence intervals will be estimated using the Clopper-Pearson method.
Percentage of subjects achieving seroconversion | Up to 180 days after immunization
  Seroconversion is defined as the percentage of subjects with either a pre-vaccination HI titer < 1:10 and a post-vaccination HI titer > 1:40 or a pre-vaccination HI titer > 1:10 and a minimum four-fold rise in post-vaccination HI antibody titer (day 0, 28). Rates of seroconversion will be calculated for each patient group, and 95% exact binomial confidence intervals will be estimated using the Clopper-Pearson method.
Cohort 2: Efficacy (immune response of COVID vaccines at least 7 days after the second dose. | Up to 365 days after immunization
  Assessments will be performed at baseline (time of enrollment), day 7 after first dose of SARS-CoV2 vaccine, day of second dose of vaccine, day 8 after second dose of vaccine, and days 90, 180, and 365.
Cohort 3: Efficacy (immune response) of COVID vaccines at least 7 days after each booster vaccine dose. | From baseline up to 365 days
  Assessments will be performed after each dose of SARS-CoV2 booster vaccine.

SECONDARY OUTCOMES:
Measurement of virus-specific serum antibody levels after vaccination | Up to 180 days after immunization
  For serum antibody responses directed against the vaccine epitopes, endpoint IgG titers after vaccination at each time point will be determined.
Measurement of virus-specific plasmablasts (PBs) after influenza vaccination | Up to 180 days after immunization
  PBs responses against influenza or SARS-CoV2 will be determined by direct ex vivo enzyme-linked immunospot (ELISPOT). Changes in the PB population will be measured to assess the timing and strength of the peak immune response to vaccination.
Measurement of virus-specific memory B-cells (MBCs) after vaccination | Up to 180 days after immunization
  The frequency of hemagglutinin (HA)-specific immunoglobulin G (IgG)-secreting MBCs per total IgG-secreting cells after vaccination will be determined. Changes in the MBC population will be measured to assess the timing and strength of the peak immune response to vaccination.
Maximum fold rise in antibody titer | Up to 180 days after immunization
  Hemagglutination inhibition assays will be used to assess the timing and strength of the peak immune response to vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Chang, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia